CLINICAL TRIAL: NCT05287763
Title: Efficacy of Collagen Sponge on Palatal Wound Healing: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Collagen Sponge on Palatal Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Peihui Ding, Deputy Chief Physician, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022(024)
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Gingival Recession; Inadequately Attached Gingiva
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gelatin Sponge (Active Comparator): The palatal wound will be protected with an absorbable gelatin sponge, which will be stabilized by non-resorbable sling sutures.
  Interventions: Procedure: Palatal soft tissue graft harvesting
- Collagen Sponge (Experimental): The palatal wound will be protected with a collagen sponge, which will be stabilized by non-resorbable sling sutures.
  Interventions: Procedure: Palatal soft tissue graft harvesting

INTERVENTIONS:
Procedure: Palatal soft tissue graft harvesting — After local anaesthesia, a horizontal incision 2 mm apically from the gingival margin will be carried out using a #15C blade. The standardized rectangular graft with a thickness of 1.5 mm will be harvested from distal aspect of canine till first molar. The graft will be lifted and separated using tissue forceps and a blade till it is free from all sides.

SUMMARY:
The aim of this study is to compare the efficacy of collagen sponge and gelatin sponge on the palatal wound healing and postoperative pain following gingival graft harvesting.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of collagen sponge and gelatin sponge on the palatal wound healing and postoperative pain following gingival graft harvesting. The included patients will be randomized into two groups. The patients in control group will be treated with gelatin sponge and those in the test group will be treated with collagen sponge. The postoperative pain will be assessed by VAS scale at day 1, 3 and 7 after surgery. Epithelialization of the palatal wound will be evaluated by hydrogen peroxide test and digital photography at 1 week postoperatively. Additionally, postoperative pain, consumption of analgesics, willingness to repeat the treatment and the existence of delayed bleeding will be recorded at 1 week. At 2 weeks, 3 weeks and 1 month after surgery, epithelialization of the palatal wound and aesthetic scores will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Clinical indications utilizing free gingival grafts or de-epithelialized gingival grafts to treat either insufficient keratinized tissue or gingival recession defects
3. Full-mouth plaque score and full-mouth bleeding score lower than 20%

Exclusion Criteria:

1. Smoking
2. Pregnancy or lactation
3. Untreated periodontal disease
4. Severe systemic conditions that contraindicate surgery (diabetes, heart disease, cancer etc.)
5. Presence of coagulation disorders (history of Haemophilia, von Wille-brand disease, or anticoagulant therapy)
6. Taking medications affecting periodontal health or healing
7. Previous surgery for a palate graft harvested from the experimental sites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
epithelialization of the palatal wound evaluated by hydrogen peroxide test | at 1 week
  The appearance of bubbles means the wound is not completely epithelialized. The result will be recorded as a dichotomous variable (yes/no).
epithelialization of the palatal wound evaluated by hydrogen peroxide test | at 2 weeks
  The appearance of bubbles means the wound is not completely epithelialized. The result will be recorded as a dichotomous variable (yes/no).
epithelialization of the palatal wound evaluated by hydrogen peroxide test | at 3 weeks
  The appearance of bubbles means the wound is not completely epithelialized. The result will be recorded as a dichotomous variable (yes/no).
epithelialization of the palatal wound evaluated by hydrogen peroxide test | at 1 month
  The appearance of bubbles means the wound is not completely epithelialized. The result will be recorded as a dichotomous variable (yes/no).
epithelialization of the palatal wound evaluated by digital photography | at 1 week
  The epithelialization of the palatal wound will be recorded as "yes" or "no" according to inspectional evaluation of surface characteristics and reflection as well as clarity and distinctness of wound outline.
epithelialization of the palatal wound evaluated by digital photography | at 2 weeks
  The epithelialization of the palatal wound will be recorded as "yes" or "no" according to inspectional evaluation of surface characteristics and reflection as well as clarity and distinctness of wound outline.
epithelialization of the palatal wound evaluated by digital photography | at 3 weeks
  The epithelialization of the palatal wound will be recorded as "yes" or "no" according to inspectional evaluation of surface characteristics and reflection as well as clarity and distinctness of wound outline.
epithelialization of the palatal wound evaluated by digital photography | at 1 month
  The epithelialization of the palatal wound will be recorded as "yes" or "no" according to inspectional evaluation of surface characteristics and reflection as well as clarity and distinctness of wound outline.

SECONDARY OUTCOMES:
postoperative pain | at day 1
  using a visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst pain imaginable)
postoperative pain | at day 3
  using a visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst pain imaginable)
postoperative pain | at day 7
  using a visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst pain imaginable)
consumption of analgesics | at 1 week
  to answer the following question: Did you take any analgesics due to the palatal pain since the procedure was completed?
willingness to repeat the treatment | at 1 week
  using a VAS ranging from 0 to 10 (0 = strong unwilling and 10 = strong willing)
the existence of delayed bleeding | at 1 week
  the occurrence of prolonged hemorrhaging during the first week
aesthetic score | at 3 weeks
  assessed by judging on the color, contour, and texture of the donor sites. The total score will vary between 0 and 6 by scoring each subject from 0 to 2 (0=inharmonious with adjacent tissue, 1=moderately harmonious with adjacent tissue and 2=very harmonious with adjacent tissue).
aesthetic score | at 1 month
  assessed by judging on the color, contour, and texture of the donor sites. The total score will vary between 0 and 6 by scoring each subject from 0 to 2 (0=inharmonious with adjacent tissue, 1=moderately harmonious with adjacent tissue and 2=very harmonious with adjacent tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Peihui Ding, Doctor, Principal Investigator — The Affiliated Stomatology Hospital of Zhejiang University School of Medicine
Locations (1):
- The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No